CLINICAL TRIAL: NCT03532724
Title: Retrospective Analysis of the Clinical Outcomes From Patient Self-management of Antivitamin K Treatment at the Hospitald de Sant Pau. ORION Study
Brief Title: Clinical Outcomes From Patient Self-management of Antivitamin K Treatment
Acronym: ORION
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ORI-2017-45
Record Dates: First submitted 2018-05-08; First posted 2018-05-22 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Self Management of Oral Anticoagulation With VKA Therapy
Keywords: Patient Self-management, Acenocoumarol, Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Patient Self-Management of VKA therapy — Trained patients check weekly the INR using a portable coagulometer an decide by themselves the dosis of VKA

SUMMARY:
ORION is a retrospective, observational, one center study to evaluate the incidence of complications (both thromboembolic and bleedings) in a cohort of patients receiving Vitamin K antagonists (VKA) under a self-management program, since 2002 at the Hospital de la Santa Creu i Sant Pau in Barcelona (Spain)

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (older than 18) under chronic VKA treatment, whom performed patient self-management for any indication of oral anticoagulation.
2. Signed informed consent

Exclusion Criteria:

1. Patients younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from atrial fibrillation, or carrying a cardiac mechanical valve prostheses, or suffering any other cardiac disease with risk of arterial embolism or with a previous venous thromboembolic event with high risk of recurrence, and receiving chronic oral anticoagulation (OA) with any VKA drug, and whom have been trained in our Unit by specialized nurses on self-management of their OA by using a portable coagulometer to weekly test the International Normalized Ratio (INR)
Sampling Method: Non-Probability Sample
Enrollment: 927 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Thromboembolic events | since 1 of july of 2002 to 30th of june of 2018
  Any documented embolic stroke, peripheral arterial embolism or venous thromboembolism
Major hemorrhagic event | since 1 of july of 2002 to 30th of june of 2018
  Any documented bleeding event grade 3 or 5 in the Bleeding Assessment Research Consortium (BARC) scale

SECONDARY OUTCOMES:
Mortality | since 1 of july of 2002 to 30th of june of 2018
  Death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Souto, MD, PhD, Principal Investigator — Hospital de la Santa creu i Sant Pau - Barcelona
Locations (1):
- Hspital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No